CLINICAL TRIAL: NCT00657319
Title: Glycaemic Control and Quality of Care in Type 2 Diabetes on NovoMix® 30 Previously Treated With Mixtard® Insulins
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1939
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — The observation is performed under normal clinical practice conditions without any additionally required diagnostic/therapeutic features. Physicians are allowed to decide the treatment regimen according to the medical standards.
  Other Names: NovoMix® 30

SUMMARY:
This observational study is conducted in Europe. The objective of this retrospective observational cohort analysis is to assess the changes of glycaemic control and quality of care in those Type 2 diabetic patients who were previously treated with Mixtard® insulins after 6 months of their switch to analog premix insulin NovoMix® 30 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 2 diabetes previously treated with BHI for at least 12 months
* Analogue premix administration for the last 6 months

Exclusion Criteria:

* Known or suspected allergy to insulin aspart
* Newly diagnosed diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with type 2 diabetes mellitus on premix insulin treatment.
Sampling Method: Probability Sample
Enrollment: 3495 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
HbA1C | 6 months

SECONDARY OUTCOMES:
General conditions (reason of switch, BMI, selected laboratory parameters, quality of care) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Budapest, Hungary

REFERENCES:
- [Result] Gerö L. Improvement in metabolic control in type 2 diabetic patients after switching from biphasic human insulin (BHI) to biphasic insulin aspart 30/70 (BIAsp 30): An observational study in Hungary. ADA American Diabetes Association 2009; Country: USA City: New Orleans
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com